CLINICAL TRIAL: NCT05536830
Title: Assessment of DeMentia Nutrition Intervention Needs Among Care Recipients and carEgivers
Acronym: ADMIRE
Status: Completed | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Heather Gibbs, Associate Professor, University of Kansas Medical Center
Other Study IDs: 148085
Record Dates: First submitted 2022-09-07; First posted 2022-09-13 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Dementia
Keywords: nutrition assessment
MeSH Terms: conditions — Dementia | interventions — Nutritional Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participant dyads: Caregivers and Care Recipients: Participants will be recruited in pairs as caregivers and care recipients. All data collected is observational in nature.
  Interventions: Other: Nutrition Status

INTERVENTIONS:
Other: Nutrition Status — Participants will be examined by a registered dietitian to assess nutrition status.

SUMMARY:
Nutrition is critical for disease prevention and brain health. Malnutrition and weight loss often affect persons with Alzheimer's dementia (PWD), worsening overall health and dementia. Informal caregivers (usually family members) perform many nutrition-related tasks as part of daily care such as food preparation and feeding. Limited research, however, suggests informal caregivers experience high rates of caregiver burden, malnutrition and low health literacy. More research is needed to uncover these and other factors that may contribute to malnutrition for both PWDs and their caregivers. Nutrition literacy, or ability to navigate nutrition information to select healthy food, may be an important caregiving factor that protects both individuals from experiencing nutritional decline. Although the NIH has increased funding to support caregiver research, caregiver interventions that include nutrition are lacking. The purpose of this study is to inform the design of a future nutrition intervention study.

ELIGIBILITY:
Inclusion Criteria:

* Person with dementia: Must be an adult of any age, diagnosed with Alzheimer's dementia or other dementia, reside at home with a family caregiver or domestic partner, and have weight records at a minimum of 2 timepoints.
* Caregiver: Must be at least 18 years old, English speaking, primary caregiver who is responsible for food planning, and no overt cognitive impairment.

Exclusion Criteria:

* Person with dementia: Frontal-temporal dementia, alcohol-related dementia, Huntington's disease, schizophrenia, manic-depressive disorder, or actively participating in nutrition intervention research.
* Caregiver: Visual impairments that prevent completing questionnaires or actively participating in nutrition intervention research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited as caregiver-patient dyads, and both must fit the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-10-25 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2024-12-08 (Actual)

PRIMARY OUTCOMES:
Nutrition status of persons with dementia | 1 month
  Nutrition status will be assessed by registered dietitians, using the Mini-Nutrition Assessment (score ranges 0 to 18) and Subjective Global Assessment (score ranges 0-7). Scores of each measure are further categorized into "normal," "at risk of malnutrition," or "malnourished."
Nutrition literacy of caregivers | 1 week
  Nutrition literacy will be measured by the Nutrition Literacy Assessment Instrument (score ranges 0 to 42). Scores are interpreted as: >39 good, 29-38: moderate, ≤ 28: poor.
Nutrition status of caregivers | 1 month
  Nutrition status of caregivers will be measured using the Mini Nutrition Assessment (MNA) tool (18-item version). Scoring is Normal (12-14 pts), At risk of malnutrition (8-11 pts), or Malnourished (0-7 points).

SECONDARY OUTCOMES:
Perceived nutrition needs of informal caregivers of persons with dementia | 1 week
  Researchers will use interviews, surveys, and focus groups to collect the thoughts of caregivers and clinic care providers to anticipate needs for a future caregiver intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Heather D Gibbs, PhD, RD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No